CLINICAL TRIAL: NCT02794662
Title: Environmental or Nasal Cannula Oxygen for Preterm Infants Receiving Oxygen Therapy: a Randomized Cross-over Pilot Study
Acronym: ECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Colm Travers, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UAB Neo 015
Record Dates: First submitted 2016-05-10; First posted 2016-06-09 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Infant, Newborn, Diseases; Hypoxia
Keywords: Oxygen Delivery System, Nasal Cannula; Oxygen Delivery System, Incubator
MeSH Terms: conditions — Infant, Newborn, Diseases; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxygen Environment (Experimental): Blended oxygen delivered by servo-controlled incubator
  Interventions: Procedure: Oxygen Environment
- Nasal cannula oxygen (Active Comparator): Blended oxygen delivered by nasal cannula
  Interventions: Procedure: Nasal Cannula Oxygen

INTERVENTIONS:
Procedure: Oxygen Environment — FiO2 delivered by servo-controlled incubator
  Arms: Oxygen Environment
Procedure: Nasal Cannula Oxygen — FiO2 delivered by nasal cannula
  Arms: Nasal cannula oxygen

SUMMARY:
The purpose of this study is to determine if, in preterm infants < 37 weeks' gestation at birth receiving oxygen without ventilatory/CPAP support, oxygen environment (OE) compared with nasal cannula oxygen (NC), will decrease the number of episodes with oxygen saturations less than 85% of ≥10 seconds in a 48 hour cross over period on either intervention.

This is a randomized cross-over pilot study with a 1:1 parallel allocation of infants to oxygen environment or nasal cannula oxygen using stratified permuted block design. Following a 24 hour period on the first intervention, infants will cross over to a 24 hour period on the second (alternative) intervention before crossing back to the first intervention for a further 24 hours and then back again to the second (alternative) intervention for a further 24 hours.

DETAILED DESCRIPTION:
In preterm infants < 37 weeks' gestation at birth requiring oxygen without ventilatory/CPAP support, will oxygen environment decrease the number of episodes with oxygen saturations less than 85% for ≥ 10 seconds in a 48 hour cross-over period on either intervention compared with nasal cannula oxygen?

The target oxygen saturations (91 to 95%) are based on data from the meta-analysis of randomized controlled trials of oxygen saturation targets which included data on 4911 infants from the SUPPORT, COT, and BOOST II trials.

This study will include preterm infants < 37 weeks' gestation on oxygen therapy via OE or NC with flow rates ≤ 1.0 l/kg/min. There will be three randomization strata [≥ 22+0/7 to ≤ 25+6/7 weeks, ≥ 26+0/7 to ≤ 28+6/7 weeks, ≥ 29+0/7 to ≤ 36+6/7 weeks' gestation]. The purpose of stratification is to ensure an appropriate distribution of risk between study arms. This study will not be powered to detect outcome differences within or between strata.

Following informed consent, randomization, stratified by gestational age at delivery, will be performed using sequentially numbered sealed opaque envelopes. Each envelope will indicate either Treatment group (OE group) or Control group (NC group). The envelope will only be opened after informed consent has been obtained and just before starting the study on each infant.

This will be a single center randomized cross-over pilot study with a 1:1 parallel allocation of infants to oxygen environment or nasal cannula oxygen using stratified permuted block design. Following a 24 hour period on the first intervention and a 15-30 minute washout period, infants will cross-over to a 24 hour period of the second/alternate intervention. Following a further 15-30 minute washout period, infants will cross-over to a 24 hour period on the first intervention. Following another 15-30 minute washout period, infants will cross-over to a 24 hour period on the second/alternate intervention. The effective FiO2 will be calculated for all infants based on their oxygen therapy modality prior to the monitoring period and used to swap between modes.

All infants enrolled in the study will have routine monitoring, uniform target saturation ranges of 91-95% with alarm limits set at 88-95%, and standard care for the duration of the study. Pulse oximetry recordings will be downloaded using ixTrend (iexcellence, Wildau, Germany) software to a secure computer system for later data analysis.

Infants will continue standard treatment as recommended by the treating physician and will act as their own controls.

Primary secondary outcomes are described below. Other safety outcomes include recordings of episodes of bradycardia and circumstances surrounding the event.

Pulse oximetry recordings will be downloaded using ixTrend software to a secure computer system for later data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Infant requiring supplemental oxygen therapy via oxygen environment (OE) or nasal cannula (NC) with flow rates ≤ 1.0 liter per kilogram per minute
* Off ventilatory support and/or NCPAP for > 48 hours prior to study entry
* Gestational age < 37 weeks' gestation at birth
* Nursed in incubator for thermoregulation
* Parents/legal guardians have provided consent for enrollment

Exclusion Criteria:

* A major malformation
* A neuromuscular condition that affects respiration
* Terminal illness or decision to withhold or limit support

Ages: 1 Hour to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The number of episodes with oxygen saturations less than 85% for ≥10 seconds | During a 48 hour cross-over period on either intervention

SECONDARY OUTCOMES:
The proportion of time with oxygen saturations > 95% | During a 48 hour cross-over period on either intervention
The coefficient of variation (relative standard deviation) of oxygen saturations | During a 48 hour cross-over period on either intervention
  The coefficient of variation is a standardized measure of dispersion of a frequency distribution defined as the ratio of the standard deviation to the mean. It will be used in this study to assess the stability of oxygen saturations.
The proportion of time spent outside oxygen saturation target ranges (91-95 %) | During a 48 hour cross-over period on either intervention
The proportion of time with oxygen saturations less than 85 % | During a 48 hour cross-over period on either intervention
The effective fraction of inspired oxygen (FiO2) requirement | During a 48 hour cross-over period on either intervention
  Effective FiO2 requirement is the actual fraction of inspired oxygen measured at the hypopharynx. In this study we will use tables based on studies where this has been previously calculated to determine the effective FiO2 requirement on the different modes of oxygen therapy during the study period.
The number of recorded interventions with tactile stimulation/blow by oxygen/CPAP/IPPV | During a 48 hour cross-over period on either intervention
  Each intervention recorded in the electronic medical record will count as 1 intervention regardless of which intervention is recorded. Therefore the same unit of measurement will be used to assess each measure.
The number of adjustments in FiO2 recorded in the electronic medical record | During a 48 hour cross-over period on either intervention
The number of episodes (≥ 10 seconds) with oxygen saturations less than 80% | During a 48 hour cross-over period on either intervention
The number of recorded episodes of bradycardia <80/min | During a 48 hour cross-over period on either intervention

CONTACTS AND LOCATIONS:
Overall Officials: Colm P Travers, MB BCh BAO, Principal Investigator — University of Alabama at Birmingham; Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Travers CP, Carlo WA, Nakhmani A, Bhatia S, Gentle SJ, Amperayani VA, Indic P, Aban I, Ambalavanan N. Environmental or Nasal Cannula Supplemental Oxygen for Preterm Infants: A Randomized Cross-Over Trial. J Pediatr. 2018 Sep;200:98-103. doi: 10.1016/j.jpeds.2018.03.010. Epub 2018 Apr 25. PMID 29705116